CLINICAL TRIAL: NCT03991689
Title: The Effect of Solution-focused Group Therapy for Pain Management in Patients With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Yu-Chan Li, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NTUNHS
Record Dates: First submitted 2019-06-09; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Pain Management; Life Quality; Spinal Cord Injuries
Keywords: spinal cord injury; pain management; pain intensity; pain self-efficacy; solution-focused group therapy
MeSH Terms: conditions — Agnosia; Spinal Cord Injuries; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the six weeks solution-focused pain management groups (Experimental)
  Interventions: Behavioral: solution-focused group therapy

INTERVENTIONS:
Behavioral: solution-focused group therapy — Participants began a 90-minute solution-focused pain management group, which lasted for six weeks, and after the group ended, the questionnaire post-test was carried out, and a total of 26 participants thus completed their group journey. The group effect was evaluated by the difference between the scores of the questionnaires before and after the group.

SUMMARY:
Objective: to verify the effect of solution-focused group therapy (SFBT) on pain management as well as physiological, psychological and social adaptation in patients with spinal cord injury.

Setting: for matters of convenience, the samples were collected at medical and rehabilitation centers in Taiwan. Twenty-six patients with spinal cord injuries and neuropathic pain were invited to join the four pain management groups.

Method: In the case of patients with spinal cord injury affected by neuropathic pain, a solution-focused pain management group therapy was conducted once a week for 6 weeks, 90 minutes each time; fear avoidance theory and acceptance and commitment therapy was used for pain management, using solution-focus group counseling strategies to guide group members to achieve pain management goals by accepting pain and establishing goals.The group effectiveness was assessed before and after the group intervention in terms of pain intensity (0-10 numeric rating scale), brief pain inventory-pain inference, chronic pain self-efficacy scale, pain fear (0-10 numeric rating scale), depression (patient health questionnaire-9), demoralization (demoralization scale), post-traumatic growth inventory and life quality (WHOQOL-BREF). Then we analyzed the correlation between the difference values of the variables before and after the test in order to understand the clinical application of the pain management group therapy for patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with spinal cord injury as being in compliance with the Taiwan National Health Insurance's definition

Exclusion Criteria:

* Psychiatric disabilities
* Intellectual disabilities
* Unconscious patients
* Patients in critical condition
* Bedridden patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04-29 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
The pain intensity and pain fear scale | 6 weeks
  The pain intensity and pain fear scale is based on the Numeric Rating Scale, asking participants "the intensity of pain in your body now" and "the degree of fear towards the future caused by your physical pain", from a minimum of 0 to a maximum of 10.
Brief Pain Inventory-Pain inference | 6 weeks
  Participants are asked to answer the extent to which pain interferes with daily life, mood, relationships with others, sleep, breathing, cough, mobility, and enjoyment of life over the past 24 hours, with a score of 0 representing no interference to 10 points representing complete interference. The total score ranges from 0 to 70, and the higher the score, the greater the degree of interference from pain.
Pain management self-efficacy subscale and symptom response self-efficacy subscale within Chronic Pain Self-Efficacy Scale (CPSS) | 6 weeks
  Since most of the patients with spinal cord injury were injured in the whole body or in the lower part of their body, the self-efficacy of their physical functions could not be revealed. Therefore, the 9 questions regarding the body function self-efficacy subscale were removed and revised into 13 questions regarding the pain self-efficacy. Participants used 0 to 10 points to indicate their degree of confidence in management and response to the situation described; 0 points indicate complete uncertainty, 10 points indicate 10% confidence, and the total score ranged from 0 to 130 points.
The depression scale uses Patient Health Questionnaires-9 | 6 weeks
  participants are asked to answer the frequency of symptoms described in the topic over the past two weeks, namely 0 points in case there were no symptoms, several days (1 point), more than one week (2 points) and almost every day (3 points) score. The total score ranges from 0 to 27 points. The higher the score, the more serious the depression.
Demoralization scale - Mandarin Version (DS-M) | 6 weeks
  DS-M includes loss of meaning, dysphoria, disheartenment, sense of failure, helplessness, and other items for total of 24 questions, with a score ranging from 0 to 4, namely from completely disagree to completely agree. The total score ranges from 0 to 96 points. The higher the score, the higher the degree of demoralization.
Post-traumatic growth inventory (PTGI) | 6 weeks
  PTGI assesses an individual's possible positive psychological changes after major stress events, including increasing the relation with others, opening up to new possibilities, increasing personal strength, appreciation of life, and spiritual change. The scale has a total of 21 questions, 0-5 points indicating a scale from no change to a very large degree of change. The total score ranges from 0 to 105 points. Spinal cord injury is mostly caused by accidents. So for a part of those with post-traumatic stress disorder (PTSD), it is estimated that post-traumatic growth can provide information about the psychological recovery of people with spinal cord injury.
The quality of life adopts Taiwan's concise version of the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF-TW) | 6 weeks
  It is made up of the 26 questions of WHOQOL-BREF , plus 2 questions related to Taiwan, for a total of 28 questions. The individual score ranges from 1 to 5. The total score ranges from 0 to 140. The higher the score, the better the quality of life.

IPD SHARING:
Plan to Share IPD: No